CLINICAL TRIAL: NCT04824261
Title: Effectiveness of 4% Boric Acid in Distilled Water Versus Clotrimazole Solution in Otomycosis Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Hosny Kamal Gendi, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: otomycosis
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): randomized 50 otomycosis patients will receive Clotrimazol solution 1%
  Interventions: Drug: Clotrimazol solution 1%
- group 2 (Active Comparator): randomized 50 otomycosis patients will receive 4%boric acid in distilled water
  Interventions: Drug: 4%boric acid in distilled water

INTERVENTIONS:
Drug: Clotrimazol solution 1% — 50 otomycosis randomized patients will receive Clotrimazol solution 1% The treatment will be locally applied for at least 2 weeks. All the patients will be followed up after the 1st week, 2nd week and after 1 month.
  Arms: group 1
Drug: 4%boric acid in distilled water — 50 otomycosis randomized patients will receive 4%boric acid in distilled water The treatment will be locally applied for at least 2 weeks. All the patients will be followed up after the 1st week, 2nd week and after 1 month.
  Arms: group 2

SUMMARY:
Otomycosis is a fungal infection that affects one, or occasionally both, of the ears. It mostly affects people who live in warm or tropical areas. It also often affects people who swim frequently, live with diabetes, or have other chronic medical and skin conditions. It is a pathologic entity, with candida and aspergillus the most common fungal species. ]Various predisposing factors include a humid climate, presence of cerumen, instrumentation of the ear, increased use of topical antibiotics / steroid preparations, immune-compromised host, patients who have undergone open cavity mastoidectomy and those who wear hearing aids with occlusive ear mold. The infection is usually unilateral and characterized by inflammatory pruritis, scaling and otalgia.Treatment recommendations have included local debridement, local and systemic antifungal agents and discontinuation of topical antibiotics. Sometimes otomycosis presents as a challenging disease for its long term treatment and follow up, yet its recurrence rate remains high.

According to Thai National List of essential medicines for topical antifugal agents are:

* acetic acid (2% in aqueous and 2% in 70% isopropyl alcohol)
* boric acid (4% in distilled water)
* gentian violet
* clotrimazole ear drop. Some fungal infections such as Aspergillus may be resistant to the usual ear drops. They may require oral medications.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic otomycosis.
* Microscopic direct examination and/or culture positive for fungus.

Exclusion Criteria:

* During usage of systemic antifungal drug
* Allergic to 4% boric acid in distilled water or clotrimazole solution

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Curative rate of otomycosis | 1 month

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ho T, Vrabec JT, Yoo D, Coker NJ. Otomycosis: clinical features and treatment implications. Otolaryngol Head Neck Surg. 2006 Nov;135(5):787-91. doi: 10.1016/j.otohns.2006.07.008. PMID 17071313
- [Background] Mugliston T, O'Donoghue G. Otomycosis--a continuing problem. J Laryngol Otol. 1985 Apr;99(4):327-33. doi: 10.1017/s002221510009678x. PMID 4009029
- [Background] Kaur R, Mittal N, Kakkar M, Aggarwal AK, Mathur MD. Otomycosis: a clinicomycologic study. Ear Nose Throat J. 2000 Aug;79(8):606-9. PMID 10969470